CLINICAL TRIAL: NCT01860911
Title: Regulation of the Plasma Triglyceride Extraction in Muscle in Insulin Resistance
Brief Title: Plasma Triglyceride Extraction by The Muscle
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Lori R. Roust, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-005173
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Insulin; omega-N-Methylarginine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin-Sensitive (Experimental): One group consists of insulin sensitive volunteers.
  Interventions: Drug: Insulin; Drug: NG-monomethyl-L-arginine
- Insulin-Resistant (Experimental): One group consists of insulin resistant volunteers.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin
Drug: NG-monomethyl-L-arginine
  Arms: Insulin-Sensitive

SUMMARY:
Increased accumulation of fat into the muscles is associated with what is called insulin-resistant state, which is a pre-diabetic state. The purpose of this research is to find out how fat circulating in the blood following fat consumption is taken up by the muscles in healthy people as well as people that are insulin-resistant. The investigators are specifically interested in how a hormone called insulin is involved in this process. Findings from this research will contribute to our understanding of why insulin-resistant people have increased accumulation of fat in their muscles, and ultimately help to design appropriate interventions to prevent type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): < 25 kg/m2 or > 30 kg/m2;
* Insulin sensitivity index (ISI): insulin-sensitive ISI ≥ 7, insulin-resistant ISI ≤ 5.

Exclusion Criteria:

* Medication or supplements known to affect either endothelial function or lipid metabolism (i.e. arginine, protein, fish oil)
* Acute illness
* Uncontrolled metabolic disease, including liver or renal disease
* Atrial fibrillation, history of syncope, limiting or unstable angina, congestive heart failure, known or suspected right-to-left, bi-directional or transient right-to-left cardiac shunts
* Cardiac pacemaker or other medical device implanted in the body
* Pulmonary hypertension or other unstable cardiopulmonary conditions
* ECG documented abnormalities or valvular disease
* Low hemoglobin or hematocrit (i.e., lower than accepted laboratory values)
* History of hypertension or elevated blood pressure (systolic, >140 mmHg or a diastolic, >95 mmHg)
* History of hyperlipidemia or plasma triglyceride concentration >200 mg/dl
* Diagnosed diabetes, or 2-h plasma glucose >200 mg/dl during an oral glucose tolerance test
* Current participation in a weight-loss regimen, including extreme dietary practices
* Use of anabolic steroids or corticosteroids (within 3 months)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Triglyceride extraction across the forearm | Measured during a 7-hour infusion study

SECONDARY OUTCOMES:
Muscle microvascular blood volume | Selected 15-minute periods during the 7 hour infusion study

CONTACTS AND LOCATIONS:
Overall Officials: Lori Roust, MD, Principal Investigator — Mayo Clinic; Christos S Katsanos, PhD, Principal Investigator — Arizona State University/Mayo Clinic Arizona
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials